CLINICAL TRIAL: NCT06900400
Title: Evaluation of Sustained Endogenous Attention Deficits in Attention Deficit Hyperactivity Disorder: Validation of a Computerized Neuropsychological Test."
Brief Title: Sustained Endogenous Attention Deficits in Attention Deficit Hyperactivity Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1064
Record Dates: First submitted 2025-03-20; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: ADHD - Attention Deficit Disorder With Hyperactivity
Keywords: Case control; diagnostic; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Disease

STUDY DESIGN:
Intervention Model Description: The same neuropsychological test is administered to two groups of subjects: one group of subjects with ADHD and one group of typically developing subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ADHD group and Control Group (Other): The same neuropsychological test (i.e.Sustained-Paced Finger Tapping) is administered to two groups of subjects: one group of subjects with ADHD and one group of typically developing subjects. Sustained-Paced Finger Tapping" (Petilli et al., 2018) is a computerized test that lasts approximately 10 minutes. It involves maintaining and reproducing the rhythm of a sound (auditory version) .
  Interventions: Diagnostic Test: Sustained-Paced Finger Tapping" (Petilli et al., 2018)

INTERVENTIONS:
Diagnostic Test: Sustained-Paced Finger Tapping" (Petilli et al., 2018) — Sustained-Paced Finger Tapping" (Petilli et al., 2018) a computerized test that lasts approximately 10 minutes. It involves maintaining and reproducing the rhythm of a sound (auditory version).

SUMMARY:
Subjects with ADHD may exhibit deficits in sustained internal attention. The "Sustained-Paced Finger Tapping" test was recently developed and experimentally used in international literature to assess sustained internal attention in typically developing children. This clinical study has several objectives: 1) to assess the presence of "internal" sustained attention deficits in children with ADHD through the "Sustained-Paced Finger Tapping"; 2) to evaluate the discriminant and ecological validity of the "Sustained-Paced Finger Tapping."

DETAILED DESCRIPTION:
Recently, a distinction has been recognized between external sustained attention and internal sustained attention. Internal sustained attention is defined as the ability to maintain attention over time on neurocognitive processes that, rather than processing external information, act on information stored in memory. The "Sustained-Paced Finger Tapping" test was developed and used in experimental research protocols in international literature to assess internal sustained attention in typically developing children. While numerous studies confirm that ADHD is associated with deficits in external sustained attention, the international literature emphasizes that internal attention has been underexplored in ADHD. A pilot study conducted by the University of Salento revealed preliminary data showing that children with ADHD exhibit significantly lower performance compared to control subjects in the "Sustained-Paced Finger Tapping." Despite these preliminary data suggesting that the "Sustained-Paced Finger Tapping" test has the ability to discriminate between children with and without ADHD, there are no published studies formally investigating this hypothesis. Two subject samples will be recruited: one sample of subjects with ADHD and one sample of subjects without ADHD and with typical development. The ADHD diagnosis will be made based on the concordance of four data sources: 1) the detection of diagnostic criteria indicated in the DSM-5 through interviews, medical history, and observation during a neuropsychiatric and psychological visit; 2) high and/or medium-high scores, i.e., ≥ 65/70 T, on the ADHD symptom subscales of both the Conners-3-Parent and the CBCL-Parent; 3) high and/or medium-high scores, i.e., ≥ 65/70 T, on the ADHD symptom subscales of at least one questionnaire (Conners-3 or CBCL) administered to teachers; 4) the presence of all DSM-5 symptoms for ADHD on the Conners-3 scale for both parents and teachers.

Inclusion criteria:

ADHD Group:

Subjects with a diagnosis of ADHD (of any severity level and subtype) aged between 6 and 10 years; "Medication-naive" ADHD subjects, i.e., subjects who have not been prescribed and/or have not yet started taking any medication for ADHD; IQ ≥ 70.

Non-ADHD Group:

Normal IQ; Aged between 6 and 10 years.

Exclusion criteria:

Exclusion criteria for both groups:

Symptoms suggestive of autism spectrum disorders, psychotic disorders, mood disorders, and anxiety disorders; Use of psychotropic drugs; Subjects with cerebral palsy and/or neuromotor and neuromuscular disorders; CNS diseases (e.g., epilepsy and/or neurodegenerative diseases) or CNS injuries due to, for example, head trauma or stroke.

The assessment of autism spectrum disorder symptoms will be carried out using the SRS-2 questionnaire, while the evaluation of other exclusion criteria will be done through medical history and clinical interview during enrollment.

Exclusion criteria for the non-ADHD group:

Presence of ADHD symptoms as identified through clinical interview and administration of a questionnaire (questionnaire from the BIA battery).

Both groups of subjects will be administered the "Sustained-Paced Finger Tapping". It is a computerized test that lasts approximately 10 minutes. It consists of maintaining and reproducing for a certain period of time (10 minutes) the rhythm of a sound presentation (auditory version).

Depending on the variables to be analyzed, non-parametric statistics or the Student's t-test and/or ANOVA will be used. ANCOVA will be employed to assess significant differences between the study variables, accounting for variables that could influence the potential differences (e.g., demographic differences between groups). ROC curve analysis, the Youden Index, and the specific formulas for calculating the diagnostic characteristics of the test will be used. The discriminant validity and the presence of any deficits in the performance related to the test will be evaluated in two ways:

1. by comparing the performances obtained from subjects with and without ADHD. To this end, the Student's t-test and/or analysis of variance (ANOVA) will be used, and if significant differences are found between the two groups regarding variables other than the dependent variables, ANCOVA will be implemented;
2. by calculating sensitivity, specificity, accuracy indices, and test cut-offs. These parameters will be calculated using the ADHD diagnosis as the gold standard for the subjects with ADHD.

The cut-off will be calculated through ROC curve analysis and the Youden Index. By "cut-off" of the test, we mean the score that best discriminates, with a certain degree of accuracy, the optimal balance between sensitivity and specificity, separating subjects with ADHD from those without ADHD. In this sense, the cut-off is considered a measure of discriminant validity, similar to statistically significant differences that can be identified using other statistical techniques.

Ecological validity will be assessed by calculating correlations and regressions between the test scores and the scores obtained on the Conners scales. Finally, simple and partial correlations will be calculated between the Sustained-Paced Finger Tapping scores and the scores from other neuropsychological tests and questionnaires administered in order to gather information on various types of validity of the instrument (construct validity, divergent, and convergent validity).

ELIGIBILITY:
Inclusion Criteria:

* ADHD Group (1) Subjects with a diagnosis of ADHD of any severity level and subtype
* ADHD Group (2) "Medication-naive" ADHD subjects, meaning subjects who have not been prescribed and/or have not yet started any pharmacological treatment for ADHD
* ADHD Group (3) IQ ≥ 70
* Non-ADHD Group, Normal IQ

Exclusion Criteria:

* for both groups, symptomatology suggestive of autism spectrum disorders, psychotic disorders, mood disorders, and anxiety disorders
* for both groups, use of psychotropic drugs
* for both groups, subjects with cerebral palsy and/or neuromotor and neuromuscular disorders
* for both groups, CNS diseases, e.g., epilepsy and/or neurodegenerative diseases, or central nervous system injuries resulting from, for example, head trauma or stroke
* for the non-ADHD group, presence of ADHD symptoms

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Performances on Sustained-Paced Finger Tapping test | baseline
  Both groups of subjects (i.e. ADHD group and Control Group) will be administered the "Sustained-Paced Finger Tapping" (Petilli et al., 2018). It is a computerized test that lasts approximately 10 minutes. It consists of maintaining and reproducing for a certain period of time (10 minutes) the rhythm of a sound presentation (auditory version).

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Associazione "La Nostra Famiglia"-IRCCS "E. Medea"-Scientific Hospital for Neurorehabilitation-Unit for Severe Disabilities in Developmental Age and Young Adults (Developmental Neurology and Neurorehabilitation), Brindisi
  - Università del Salento, Lecce